CLINICAL TRIAL: NCT03483402
Title: Study of the Efficacy of a Single Session Micropulse Laser Trabeculoplasty as an Adjunctive Measure in Decreasing Intraocular Pressure in Patients Suffering From Pseudoexfoliation Glaucoma
Brief Title: Micropulse Laser Trabeculoplasty as Adjunctive Treatment in Patients With Pseudoexfoliation Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Constantinos D. Georgakopoulos, MD, PhD, Associate Professor in Ophthalmology, University Hospital of Patras
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 58/15.02.2018/5103
Record Dates: First submitted 2018-03-23; First posted 2018-03-30 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Pseudoexfoliation Glaucoma; Primary Open-angle Glaucoma
Keywords: Pseudoexfoliation Glaucoma; Primary Open-angle Glaucoma; Micropulse Laser Trabeculoplasty; Intraocular Pressure
MeSH Terms: conditions — Exfoliation Syndrome; Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: Single-center, one-arm, prospective clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEXG treated with MLT (Experimental): Patients with pseudoexfoliation glaucoma (PEXG) under prostaglandine analogue monotherapy with inadequate IOP control treated with 360-degrees 532nm micropulse laser trabeculoplasty (MLT)
  Interventions: Procedure: Micropulse laser trabeculoplasty

INTERVENTIONS:
Procedure: Micropulse laser trabeculoplasty — Micropulse laser trabeculoplasty is performed using the Iridex IQ 532 laser system (Iridex Corporation, 1212 Terra Bella Avenue, Mountain View, CA, USA) and 532 nm (green) wavelength MLT is applied with confluent applications to pigmented trabecular meshwork over 360 degrees using a 300 µm spot size, 300 ms duration, 1000 mW power and 15% duty cycle.
  Other Names: MLT Iridex IQ 532 laser system

SUMMARY:
This study aims to evaluate the effect of a single session of micropulse laser trabeculoplasty (MLT) on cornea in eyes with primary open glaucoma (POAG) and pseudoexfoliation glaucoma (PEXG).

DETAILED DESCRIPTION:
Patients with PEXG under prostaglandine analogue monotherapy with inadequate IOP control are treated with 360-degrees 532nm MLT.

Patients are evaluated at 1 day, 1 month, 3 months, 6 months and 12 months post-MLT. After trabeculoplasty patients are maintained in treatment with the same drug regimen as pre-MLT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with POAG or PEXG under treatment with glaucoma agents requiring additional reduction of IOP, age older than 18 years, patients willing to provide informed consent to participate in the study and to adhere to the follow-up schedule.

Exclusion Criteria:

* pre-existing corneal pathology or scar, history of any previous ocular surgery or any planned ocular surgery during the study, history of prior laser trabeculoplasty, end-stage glaucoma with advanced visual field defect, monocular patients, history of trauma, and concurrent systemic or topical steroid use
* patients unable to present for follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure | 12 months
  The change in IOP at 12 months versus baseline and the percentage of patients with ≥20% reduction in IOP.

SECONDARY OUTCOMES:
Intraocular Pressure | 1, 3 and 6 months
  Change in IOP and the percentage of ≥20% IOP reduction at 1, 3 and 6 months after MLT

CONTACTS AND LOCATIONS:
Overall Officials: Constantine D Georgakopoulos, MD, PhD, Principal Investigator — University of Patras, Medical School

REFERENCES:
- [Derived] Makri OE, Pallikari A, Pagoulatos D, Kagkelaris K, Kostopoulou EV, Georgakopoulos CD. Micropulse laser trabeculoplasty on pseuodexfoliation glaucoma patients under topical prostaglandin analogue monotherapy: 1-year results. Graefes Arch Clin Exp Ophthalmol. 2019 Feb;257(2):349-355. doi: 10.1007/s00417-018-4195-2. Epub 2018 Nov 28. PMID 30488265